CLINICAL TRIAL: NCT00505232
Title: Induction Treatment With Anti-CD20 Plus Hyper-CVAD and Methotrexate/Cytarabine Followed by Consolidation Treatment With Y90 Ibritumomab-Tiuxetan in Patients With Mantle Cell Lymphoma
Brief Title: Safety Study to Evaluate Induction and Consolidation Treatment in Patients With Mantle Cell Lymphoma (LCM-04-02)
Acronym: LCM-04-02
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CABYC (Industry)
Collaborators: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GELTAMO-LCM-04-02; 2005-004400-37 (EudraCT Number)
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2012-01-02 (Estimated); Status verified 2011-12

CONDITIONS: Mantle Cell Lymphoma
Keywords: Y-90 Ibritumomab tiuxetan; Rituximab; Hyper-CVAD; Mantle Cell Lymphoma Patients; Zevalin(R)
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab-HCVAD,Methotrexate/Cytarabine and Zevalin (Experimental): Induction Treatment (Rituximab-HCVAD and Methotrexate/Cytarabine) followed by Consolidation Treatment (Rituximab and Y-90 Ibritumomab tiuxetan)
  Interventions: Drug: Y-90 Ibritumomab tiuxetan

INTERVENTIONS:
Drug: Y-90 Ibritumomab tiuxetan — Study Design
  The present study will be split into two cohorts:
  1. Patients younger than 60 years who will receive 8 chemotherapy cycles
  2. Patients older than 60 years who will receive 6 chemotherapy cycles
  The induction schema summarises as follows :
  Anti-CD20/Hyper -CVAD chemotherapy will be alternated with anti-CD20 +MTX/Ara-C chemotherapy twice. Afterward, response will be evaluated, followed by, either, four cycles further patients younger than 60 years who will obtain a CR or PR, or 2 cycles patients older than 60 y. (see figure 1 and flow chart).
  Consolidation treatment will consist in a single dose of Y90-Ibritumomab -Tiuxetan (Zevalin) [0.4 mCi/Kg b.w or 0.3 mCi/kg if platelets < 100,000/µl] will be administered 8 to 12 weeks after last chemotherapy.

SUMMARY:
Mantle Cell Lymphoma (MCL) is a malignancy with a poor response to treatment and with a median survival of 2- 4 years since diagnosis. Although histology is similar to that of an indolent lymphoma, MCL is currently considered an aggressive tumour. Few prospective therapeutic trials have been reported in MCL, and results are difficult to interpret due to treatment heterogeneity. It is known that standard chemotherapy for other clinically aggressive lymphomas yields poor results. Recently, better results have been communicated with intense induction chemotherapy treatments or consolidating the response with high dose chemotherapy with stem cell support. Keeping in mind these considerations, we will use and intensive induction treatment with Hyper-CVAD/MTX-AraC associated with anti-CD20 in order to increase the overall response rate followed by consolidation treatment with Ibritumomab -tiuxetan (Zevalin) with the aim of eradicate the minimal residual disease, responsible of relapse.

DETAILED DESCRIPTION:
Study Design:

* The Patients will receive 6 cycles of induction chemotherapy as follows: Anti-CD20/Hyper -CVAD chemotherapy will be alternated with anti-CD20 +MTX/Ara-C chemotherapy. After 4 cycles (2 x2), response will be evaluated. If response (complete or partial) is observed, 2 additional cycles will be administrated. If less than a partial response is observed, the patient will be out of the study.
* Consolidation treatment will be a single dose of Y90Ibritumomab -Tiuxetan (Zevalin) will be administered after 12 weeks after completion of induction chemotherapy. The initial dose of Zevalin will be 0.3 mCi/kg, to be further escalated to 0.4 mCi/Kg if unacceptable toxicity does not occur.

ELIGIBILITY:
Inclusion Criteria:

* All histologic MCL subtypes (WHO classification)
* Age between 18 and 70 years old
* Performance status 0 to 2 (ECOG)
* Cardiac ejection fraction >50%
* Adequate organ (hepatic, cardiac and renal) and marrow function: Hb> 10g/dl, neutrophil counts> 1500/ µl, platelet> 100000/ µl. Creatinine < 2,5xULN, bilirubin, AST or ALT<2,5xULN.
* For Y90-ibritumomab tiuxetan administration: Bone Marrow Infiltration by lymphoma cells < than 25% ; platelet count >100,000/µl and neutrophil counts >1500/µl
* Informed consent should be obtained

Exclusion Criteria:

* Ann Arbor stages I or II without B symptoms or bulky disease (>10 cm).
* Previous chemotherapy or radiotherapy treatment.
* Uncontrolled current illness: Hepatic, renal, cardiovascular, neurological or metabolic illness.
* Symptomatic congestive heart failure, unstable angina pectoris, clinically significant cardiac arrhythmia.
* HIV, HBV or HCV positive serology.
* Limitation of the patient´s ability to comply with the treatment or follow-up protocol.
* Men and women with reproductive potential who are not using effective contraceptive methods during and at least 12 months after the end of the study
* Acute or chronic active infection.
* Known hypersensitivity to some of the drugs or other related compounds
* No informed consent obtained

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2006-01; Primary Completion 2010-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Treatment safety | 36 months
  Safety of the treatment, recording the adverse events throughout the treatment.

SECONDARY OUTCOMES:
Feasibility of proposed treatment scheme. | 36 months
  Number and percentage of patients susceptible of receiving consolidation treatment after induction chemotherapy, according to inclusion criteria for consolidation with radioinmunotherapy.
Efficacy based on response rate: overall, partial and complete response. | 36 months
Progression free, disease free and overall survivals. | 36 months
Analysis of the significance of the minimal residual disease (MRD) detection. | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Reyes Arranz, MD, PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (16):
- Spain (16):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Marques de Valdecilla, Santander, Cantabria
  - Hospital del Mar, Barcelona, Catalonia
  - Hospital Clínico de Santiago de Compostela, Santiago de Compostela, Galica
  - Clinica Ruber, Madrid, Madrid
  - Hospital La Princesa, Madrid, Madrid
  - Clinica Moncloa, Madrid, Madrid
  - Hospital Ramon y Cajal, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid, Madrid
  - Hospital Universitario La Paz, Madrid, Madrid
  - Hospital Quiron, Madrid, Madrid
  - Hospital Morales Meseguer, Murcia, Murcia
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Clínico de Salamanca, Salamanca, Salamanca
  - Hospital Clinico de Valencia, Valencia, Valencia
  - Hospital Dr. Peset, Valencia, Valencia